CLINICAL TRIAL: NCT00871169
Title: INST 0802: Phase II Trial of Combination Irinotecan, Oxaliplatin and Cetuximab for Patients With Locally Advanced or Metastatic Pancreatic Cancer
Brief Title: Combination of Irinotecan, Oxaliplatin and Cetuximab for Locally Advanced or Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New Mexico Cancer Research Alliance (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INST 0802; NCI-2011-02731 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-03-26; First posted 2009-03-30 (Estimated); Results first posted 2016-06-14 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-05

CONDITIONS: Pancreatic Cancer
Keywords: Irinotecan; Oxaliplatin; Cetuximab; Advanced or metastatic pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Irinotecan; Oxaliplatin; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Irinotecan, oxaliplatin, and cetuximab (Experimental): The goal is to administer at least 4 cycles to each patient, but treatment may stop earlier if the treating physician deems stopping to be in the best interest of the patient. Repeated treatment may be given to patients who benefit (either complete or partial response or stabilization of disease)
  Interventions: Drug: Irinotecan, oxaliplatin, and cetuximab

INTERVENTIONS:
Drug: Irinotecan, oxaliplatin, and cetuximab — Irinotecan at 90 mg/m2 intravenously every two weeks (administered over 60 minutes) + Oxaliplatin at 60 mg/m2 intravenously every two weeks(administered over 60 minutes) + Cetuximab at 250 mg/m2 intravenously every two weeks (administered over 90 minutes).
  The treatment interval (one cycle) is every 14 days.
  Other Names: Eloxatin; ERBITUX

SUMMARY:
This phase II trial studies the side effects and how well irinotecan hydrochloride, oxaliplatin and cetuximab work in treating patients with unresectable or metastatic pancreatic cancer. Irinotecan hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving irinotecan hydrochloride together with oxaliplatin and cetuximab may kill more tumor cells.

DETAILED DESCRIPTION:
The investigators will evaluate the side effects and how well irinotecan hydrochloride, oxaliplatin and cetuximab work in treating patients with unresectable or metastatic pancreatic cancer. Irinotecan hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving irinotecan hydrochloride together with oxaliplatin and cetuximab may kill more tumor cells.

ELIGIBILITY:
Inclusion Criteria:

1. All patients, 18 years of age or older, with histology proven pancreatic cancer are eligible.
2. Patients must have a life expectancy of at least 12 weeks.
3. Patients must have a Zubrod performance status of 0-2.
4. Patients must sign an informed consent.
5. Patients should have adequate bone marrow function defined by an absolute peripheral granulocyte count of >= 1,500 or cells/mm3 and platelet count >= 60,000/mm3 and absence of a regular red blood cell transfusion requirement.
6. Patients should have adequate hepatic function with a total bilirubin <= 4.0 mg/dl, could be <= 10 mg/ml if biliary drainage tube is placed and functional in a newly diagnosed patient, and SGOT or SGPT <= four times the upper limit of normal, and adequate renal function as defined by a serum creatinine <= 1.5 x upper limit of normal.
7. For patients that had been treated with one of the study medications will be allowed as long as the treatment did not contain more than 2 study medications at the same time. For example, irinotecan and capecitabine combination will be allowed but not irinotecan and cetuximab. Similarly, gemcitabine with cetuximab will be allowed but not gemcitabine, oxaliplatin and cetuximab. Treated with irinotecan alone followed by oxaliplatin will be allowed but not when irinotecan was in combination with oxaliplatin.
8. Patients are allowed to have up to 2 prior treatments. The protocol will also include chemotherapy naïve patients.

Exclusion Criteria:

1. Patients with symptomatic brain metastases are excluded from this study.
2. Pregnant women or nursing mothers are not eligible for this trial. Patients of child bearing potential must use adequate contraception.
3. Patients may receive no other concurrent chemotherapy or radiation therapy during this trial.
4. Patients with severe medical problems such as uncontrolled diabetes mellitus or cardiovascular disease or active infections are not eligible for this trial.
5. Known hypersensitivity reaction to any of the study medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2008-10; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fa-Chyi Lee, M.D., Principal Investigator — University of New Mexico Cancer Center
Locations (5):
- United States (5):
  - University of New Mexico Cancer Center @ Lovelace Medical Center, Albuquerque, New Mexico
  - Hematology Oncology Associates, Albuquerque, New Mexico
  - Cancer Center at Presbyterian Hospital, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Memorial Medical Center- Cancer Center, Las Cruces, New Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of New Mexico Cancer Center — http://www.cancer.unm.edu
- See also: New Mexico Cancer Care Alliance — http://www.nmcca.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at the University of New Mexico Comprehensive Cancer Center between October, 2008, and December, 2014.
Groups:
- Irinotecan, Oxaliplatin, and Cetuximab: The goal is to administer at least 4 cycles to each patient, but treatment may stop earlier if the treating physician deems stopping to be in the best interest of the patient. Repeated treatment may be given to patients who benefit (either complete or partial response or stabilization of disease)
  Irinotecan, oxaliplatin, and cetuximab: Irinotecan at 90 mg/m2 intravenously every two weeks (administered over 60 minutes) + Oxaliplatin at 60 mg/m2 intravenously every two weeks(administered over 60 minutes) + Cetuximab at 250 mg/m2 intravenously every two weeks (administered over 90 minutes).
  The treatment interval (one cycle) is every 14 days.
Period: Overall Study
Arm/Group | Irinotecan, Oxaliplatin, and Cetuximab
Started | 61
Completed | 58
Not Completed | 3
Not completed — Protocol Violation | 1
Not completed — Patient did not receive study treatment | 2

BASELINE CHARACTERISTICS:
Population: These enrolled patients received study treatment according to the protocol.
Arm/Group | Irinotecan, Oxaliplatin, and Cetuximab
Number analyzed (Participants) | 58
Age, Continuous [Median (Full Range); unit: years] | 62 [39 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22
  Not Hispanic or Latino | 35
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 58

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: ORR is evaluated according to Response Evaluation Criteria in Solid Tumors (RECIST) (version 1.1). Target lesions are assessed by computerized tomography (CT): Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), neither sufficient decrease in the sum of the longest diameter of target lesions to qualify for PR nor sufficient increase in the sum of the longest diameter of target lesions to qualify for Progressive Disease; Progressive Disease (PD), 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. ORR is the percentage of patients who experienced a CR + the percentage of patients who experienced a PR.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Irinotecan, Oxaliplatin, and Cetuximab
Number analyzed (Participants) | 58
percentage of participants | 6.9 [1.91 to 16.7]

2. Secondary Outcome: Toxicity
Description: Toxicity will be evaluated per National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE), version 3.0. Frequency and severity of adverse events will be tabulated using counts of frequently occurring, serious and severe events of interest (i.e. Grade 3 and Grade 4 adverse events, and Serious Adverse Events (SAEs)).
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Irinotecan, Oxaliplatin, and Cetuximab
Number analyzed (Participants) | 58
participants
  Grade 3 Alkaline Phosphatase Increased | 4
  Grade 3 Allergic Reaction/Hypersensitivity | 1
  Grade 3 Anorexia | 2
  Grade 3 Ascites | 2
  Grade 3 Aspartate Aminotransferase Increased | 1
  Grade 3 Constipation | 3
  Grade 3 Creatinine Increased | 1
  Grade 3 Hemoglobin Decreased | 2
  Grade 3 Dehydration | 1
  Grade 3 Diarrhea | 1
  Grade 3 Limb Edema | 1
  Grade 3 Fatigue | 8
  Grade 3 Gamma-glutamyltransferase Increased | 2
  Grade 3 Hyperbilirubinemia | 3
  Grade 3 Hyperglycemia | 6
  Grade 3 Hypoalbuminemia | 1
  Grade 3 Hypokalemia | 11
  Grade 3 Hyponatremia | 1
  Grade 3 Hypophosphatemia | 3
  Grade 3 Insomnia | 1
  Grade 3 Leukopenia | 1
  Grade 3 Nausea | 3
  Grade 3 Neutropenia | 3
  Grade 3 Pain - Abdomen | 5
  Grade 3 Pain - Bone | 1
  Grade 3 Decreased Respiration | 1
  Grade 3 Rash | 3
  Grade 3 Syncope | 1
  Grade 3 Thrombocytopenia | 2
  Grade 3 Vomiting | 2
  Grade 4 Encephalopathy | 1
  Grade 4 Fatigue | 1
  Grade 4 Gamma-glutamyltransferase Increased | 1
  Grade 4 Hyperglycemia | 1
  Grade 4 Hypokalemia | 1
  Grade 4 Hypothermia | 1
  Grade 4 Pleural Effusion | 1
  SAE: Grade 3 Acidosis | 1
  SAE: Grade 3 Anorexia | 1
  SAE: Grade 3 Ascites | 1
  SAE: Grade 3 Bacteremia | 1
  SAE: Grade 3 Cholangitis | 1
  SAE: Grade 3 Dehydration | 7
  SAE: Grade 3 Diarrhea | 1
  SAE: Grade 3 Fatigue | 1
  SAE: Grade 3 Gastrointestinal Hemorrhage | 2
  SAE: Grade 4 Hyperbilirubinemai | 1
  SAE: Grade 4 Hyperglycemia | 1
  SAE: Grade 3 Hypotension | 1
  SAE: Grade 2 Bowel Obstruction | 1
  SAE: Grade 3 Bowel Obstruction | 2
  SAE: Grade 3 Gholangitis | 1
  SAE: Grade 2 Urinary Tract Infection | 1
  SAE: Grade 3 Infection of unknown origin | 1
  SAE: Grade 5 Intracranial Hemorrhage | 1
  SAE: Grade 2 Mental Status Change | 1
  SAE: Grade 4 Muscle Weakness | 1
  SAE: Grade 3 Nausea | 1
  SAE: Grade 2 Abdominal Pain | 1
  SAE: Grade 3 Abdominal Pain | 4
  SAE: Grade 2 Pulmonary embolus | 1
  SAE: Grade 4 Pulmonary Embolus | 2
  SAE: Grade 4 Renal Failure | 1
  SAE: Grade 4 Seizure | 1
  SAE: Grade 2 Sinus tachycardia | 1
  SAE: Grade 4 Thrombosis | 1
  SAE: Grade 3 Vomiting | 3
  SAE: Grade 3 Weight Loss | 1

ADVERSE EVENTS:
Description: Study participants were assessed for toxicity at every scheduled study visit through a full clinical exam. Patient-reported toxicities were also collected.
Arm/Group | Irinotecan, Oxaliplatin, and Cetuximab
Serious Adverse Events (participants affected / at risk) | 24/58
Other Adverse Events (participants affected / at risk) | 56/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Irinotecan, Oxaliplatin, and Cetuximab (N=58)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Bacteremia (Infections and infestations) | 1 (1)
Cholangitis (Biliary tract infection) (Infections and infestations) | 1 (1)
Dehydration (General disorders) | 5 (7)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Hemorrhage - Gastrointestinal (Vascular disorders) | 1 (2)
Hyperbilirubinemia (Elevated bilirubin) (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (High blood glucose) (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1)
Ileus (bowel obstruction) (Gastrointestinal disorders) | 3 (3)
Infection - biliary tract (cholangitis) (Infections and infestations) | 1 (1)
Infection - Urinary tract (Infections and infestations) | 1 (1)
Infection of unknown origin (Infections and infestations) | 1 (1)
Intracranial hemorrhage (Vascular disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Pain - Abdomen (General disorders) | 5 (5)
Pulmonary Emboli (Vascular disorders) | 3 (3)
Renal failure (Renal and urinary disorders) | 1 (1)
Seizure (Psychiatric disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Thrombosis/embolism (vascular access) (Vascular disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3)
Weight loss (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Irinotecan, Oxaliplatin, and Cetuximab (N=58)
Abdominal distention (Gastrointestinal disorders) | 5 (6)
Acneiform rash (Skin and subcutaneous tissue disorders) | 5 (5)
Alanine aminotransferase increased (Metabolism and nutrition disorders) | 4 (6)
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 11 (14)
Alopecia (Skin and subcutaneous tissue disorders) | 9 (11)
Anemia (Blood and lymphatic system disorders) | 4 (5)
Anorexia (Gastrointestinal disorders) | 22 (27)
Anxiety (Nervous system disorders) | 4 (5)
Ascites (Gastrointestinal disorders) | 4 (6)
Aspartate aminotransferase increased (Metabolism and nutrition disorders) | 5 (6)
Constipation (Gastrointestinal disorders) | 18 (23)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Decreased hemoglobin (Blood and lymphatic system disorders) | 11 (18)
Dehydration (General disorders) | 6 (6)
Depression (Nervous system disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 27 (43)
Dizziness (Nervous system disorders) | 5 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 9 (9)
Dyspepsia (Heartburn) (Gastrointestinal disorders) | 5 (5)
Dyspnea (Shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Edema - limbs (General disorders) | 9 (10)
Fatigue (General disorders) | 29 (53)
Fever (General disorders) | 6 (9)
Gamma-glutamyltransferase increased (Metabolism and nutrition disorders) | 8 (11)
Hemorrhage - Nasal (Vascular disorders) | 3 (3)
Hyperbilirubinemia (High bilirubin levels) (Metabolism and nutrition disorders) | 6 (9)
Hyperglycemia (High glucose levels) (Metabolism and nutrition disorders) | 12 (25)
Hypoalbuminemia (Low blood albumin) (Metabolism and nutrition disorders) | 12 (18)
Hypocalcemia (Low calcium levels) (Metabolism and nutrition disorders) | 10 (12)
Hypokalemia (Low potassium levels) (Metabolism and nutrition disorders) | 17 (35)
Hypomagnesemia (Low magnesium levels) (Metabolism and nutrition disorders) | 7 (11)
Hyponatremia (Low sodium levels) (Metabolism and nutrition disorders) | 6 (8)
Hypophosphatemia (Low phosphate levels) (Metabolism and nutrition disorders) | 4 (10)
Infection - Urinary tract (Infections and infestations) | 3 (3)
Insomnia (Nervous system disorders) | 8 (10)
Leukopenia (Decreased leukocytes) (Blood and lymphatic system disorders) | 6 (10)
Mucositis (Gastrointestinal disorders) | 6 (7)
Nausea (Gastrointestinal disorders) | 34 (56)
Neutropenia (Decreased neutrophils) (Blood and lymphatic system disorders) | 16 (24)
Pain - Abdomen (General disorders) | 19 (32)
Pain - Back (General disorders) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 16 (22)
Pruritis (Itching) (Skin and subcutaneous tissue disorders) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 30 (44)
Rigors/chills (General disorders) | 4 (4)
Taste alteration (Gastrointestinal disorders) | 6 (7)
Thrombocytopenia (decreased platelets) (Blood and lymphatic system disorders) | 8 (14)
Vomiting (Gastrointestinal disorders) | 24 (40)
Weight loss (General disorders) | 20 (25)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No